CLINICAL TRIAL: NCT05490927
Title: Latinx Smokers: Evaluating Ethnic Microaggressions on Smoking Behavior and Relapse
Brief Title: Ethnic Microaggressions and Smoking Behaviors Among Latinx Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Brooke Kauffman, Research Assistant Professor, University of Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00003689
Record Dates: First submitted 2022-06-17; First posted 2022-08-08 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Smoking; Discrimination, Racial
Keywords: Smoking; Hispanic; Latinx
MeSH Terms: conditions — Smoking; Racism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoking Deprivation (Experimental): 16 hours of smoking abstinence prior to experimental visit.
  Interventions: Behavioral: Microaggression Recall and Relapse Analogue Task
- Smoking as Usual (Experimental): Smoking as usual prior to experimental visit.
  Interventions: Behavioral: Microaggression Recall and Relapse Analogue Task

INTERVENTIONS:
Behavioral: Microaggression Recall and Relapse Analogue Task — Participants will engage in a microaggression recall task followed by the McKee Experimental Relapse Analogue Task

SUMMARY:
The purpose of this study is to examine whether microaggressions relate to multimodal facets of smoking behavior, subjective withdrawal, and urge/craving. Additionally, the second aim is to examine whether smoking deprivation moderates the relation between microaggressions and multiple facets of smoking behavior, subjective withdrawal, and urge/craving.

DETAILED DESCRIPTION:
This proposal will employ a novel multi-modal approach to evaluate the role of microaggressions in relation to smoking lapse and topography among a sample of Latinx smokers. Adult Latinx daily smokers will attend two counterbalanced experimental sessions - (1) smoking deprivation (16 hours of smoking abstinence) and (2) smoking as usual - during which microaggressions during the relapse analog task will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Current regular (daily) cigarette smoking for >= 1 year
* Current smoking >= 5 cig/day and biochemically confirmed via carbon monoxide (CO) analysis
* Being self-identified as Hispanic or Latino
* Able to provide written, informed consent
* Endorsement of at least one microaggression experience over the past 6-months

Exclusion Criteria:

* Endorsement of current psychotic symptoms
* Active suicidality
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Smoking Behaviors | During the Smoking as Usual Visit and Smoking Deprivation Visit (Visits are randomly ordered, counterbalanced separated by ~14 days)
  Smoking behaviors will be operationally defined as smoking topography (e.g., puff behavior) measured via the Clinical Research Support System (CReSS; Plowshare Technologies, Borgwaldt KC, Inc., Virginia).
Subjective Withdrawal | During the Smoking as Usual Visit and Smoking Deprivation Visit (Visits are randomly ordered, counterbalanced separated by ~14 days)
  The 8-item Minnesota Withdrawal Scale will be used to assesses withdrawal severity. Each of the items are rated on a Likert-type scale ranging from 0 to 4. Items are summed to produce a total score with higher scores indicative of worse outcomes (possible range 0-32).
Urge/Craving | During the Smoking as Usual Visit and Smoking Deprivation Visit (Visits are randomly ordered, counterbalanced separated by ~14 days)
  Smoking urge/craving will be measured with the 10-item Questionnaire of Smoking Urges-Brief (QSU-B). Each of the items are rated on a Likert-type scale ranging from 1 to 7. Items are summed to create two subscale scores and a total score with higher scores indicative of worse outcomes (possible range 7-70).
Smoking Lapse Behaviors | During the Smoking as Usual Visit and Smoking Deprivation Visit (Visits are randomly ordered, counterbalanced separated by ~14 days)
  Smoking Lapse Behaviors will be measured during the Relapse Analogue Task (RAT), during which participants are able to delay smoking for a small financial reward. For this task, Smoking Lapse Behaviors are conceptualized as two variables: (a) minutes in time of smoking delay (possible range -50 to +50) and (b) number of cigarettes smoked

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Y Kauffman, Ph.D., Principal Investigator — University of Houston
Locations (1):
- RESTORE Laboratory: Research on Emotion, Substance Treatment Outcomes, and Racial Equity, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No